CLINICAL TRIAL: NCT02552225
Title: Double-blind Placebo Controlled Trial of the Treatment of Chronic Laryngitis With Amitriptyline
Brief Title: Treatment of Chronic Laryngitis With Amitriptyline
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding was not obtained so the study could not be continued after the Covid pause.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H 34438
Record Dates: First submitted 2015-09-09; First posted 2015-09-17 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Laryngeal Diseases
Keywords: laryngeal sensory neuropathy, chronic laryngeal neuropathy
MeSH Terms: conditions — Laryngeal Diseases | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- amitriptyline (Experimental): Subjects in this arm will receive pills composed of amitriptyline and Avicel (cellulose filler)
  Interventions: Drug: Amitriptyline
- placebo (Placebo Comparator): Subjects in this arm will receive pills composed only of Avicel (cellulose filler)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amitriptyline — Subjects in this arm will receive pills composed of amitriptyline and Avicel (cellulose filler)
  Other Names: Elavil
  Arms: amitriptyline
Other: Placebo — Subjects in this arm will receive pills composed only of Avicel (cellulose filler)
  Arms: placebo

SUMMARY:
This randomized, double-blind, placebo-controlled trial will compare the effectiveness of amitriptyline versus placebo (inactive medication) in treating chronic laryngitis.

DETAILED DESCRIPTION:
Chronic laryngitis commonly manifests through symptoms including cough, hoarseness, throat clearing, foreign body sensation, throat pain, sensation of excessive phlegm, and difficulty swallowing. A significant minority also present with GERD, rhinosinusitis-induced post-nasal drainage, direct allergic effect, and smoking issues.

Amitriptyline is commonly used for mental/mood problems, but is also prescribed to treat chronic laryngitis because some investigators suggest a neuropathic etiology for idiopathic chronic laryngitis. No trials have compared any treatment for chronic laryngitis to placebo and it is unknown if currently used therapies for chronic laryngitis are effective.

At the baseline visit, subjects will be assigned at random to amitriptyline or placebo, which they will take for 4 weeks each. Subjects will be seen in the clinic at baseline and after 10 weeks. Improvement will be measured using standardized symptom scales, and a self-reported subjective improvement percentage.

ELIGIBILITY:
Inclusion Criteria:

1. Must be age 18 or older and able to consent for themselves
2. Must have had structural pathology such as tumor previously ruled out using flexible laryngoscopy
3. Must be able to speak and read the English language
4. Must have failed a 2 month or longer trial of a proton pump inhibitor for the treatment of gastro-esophageal reflux
5. Women under 55 years of age who may become pregnant must have a negative pregnancy test and agree to barrier or hormonal methods of contraception during the study
6. Potential subject and their physician have agreed that amitriptyline will be part of their regular care plan

Exclusion Criteria:

1. Active untreated environmental allergies
2. Smoking within past 5 years
3. Current upper respiratory infections
4. Use of narcotics (e.g. oxycodone, methadone) within the past week
5. Hypersensitivity to amitriptyline
6. History of amitriptyline use or of other tricyclic antidepressant - including pregabalin, gabapentin, baclofen, or other gamma-aminobutyric acid (GABA)analogues or inhibitors - for any medical condition (not limited to chronic laryngitis) within the past 12 months.
7. Use of any other monoamine oxidase inhibitors (MAOIs) other than amitriptyline within the past 4 weeks (selegiline, phenelzine, tranylcypromine, isocarboxazid, rasagiline, phenelzine sulfate, selegiline hydrochloride, rasagiline mesylate, tranylcypromine sulfate)
8. History of urinary retention
9. History of an acute episode of a major depressive disorder within the past 12 months
10. For women 18-55 years of age without history of menopause: currently nursing or pregnant, plans to become pregnant, or unwillingness to utilize contraception (barrier or hormonal methods)
11. Currently participating in another clinical trial that could interfere with the efficacy of, or participation in, this study.
12. Current untreated diagnosis of gastroesophageal reflux (GERD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Pieter Noordzij, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amitriptyline | Placebo
Started | 3 | 3
Completed | 2 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (19.9) | 55.0 (6.6) | 53.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 2 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Reflux Symptom Index (RSI) [Mean (Standard Deviation); unit: score on a scale] — The Reflux Symptom Index (RSI) is a validated questionnaire consisting of 9 statements to be ranked on a scale of 0-5 (0=no problem, 5=severe problem). RSI scores can range from 0 to 45 with higher scores correlated with more reflux symptoms.
  score on a scale | 21.33 (11.50) | 25.67 (6.51) | 23.50 (8.69)
Voice Handicap Index-10 (VHI-10) [Mean (Standard Deviation); unit: units on a scale] — The Voice Handicap Index-10 (VHI-10) is a 10-question scale rated from 0-4 that addresses effects on quality of life from voice disorders (0=never, 1=almost never, 2=sometimes, 3=almost always, 4=always). VHI-10 scores can range from 0 to 40, with lower scores correlated with a higher quality of life related to voice disorders.
  units on a scale | 1.67 (2.89) | 9.67 (9.5) | 5.67 (7.66)
Cough Severity Index (CSI) [Mean (Standard Deviation); unit: units on a scale] — The Cough Severity Index is a validated 10 item questionnaire to quantify a patient's symptoms associated with upper airway chronic cough. The 4 point Likert scale for each of the 10 items is 0 to 4 where 0 = Never, 1 = Almost never, 2 = Sometimes, 3 = Almost always, 4 = Always. Scores can range from 0 to 40 and higher scores reflect more coughing.
  units on a scale | 4.00 (5.66) | 21.33 (12.42) | 14.40 (13.24)
Throat pain/burning [Mean (Standard Deviation); unit: units on a scale] — Participants will be asked to rate the severity of their "throat pain or burning" on a scale from 0 (no problem) to 5 (severe). Higher scores are correlated with more throat pain/burning.
  units on a scale | 0.0 (0.0) | 3.33 (1.53) | 1.67 (2.07)
Pain when swallowing [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to rate their pain when swallowing on a scale of 0=none to 5= severe pain.
  units on a scale | 0.67 (1.15) | 0.67 (0.58) | 0.67 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Reflux Symptom Index (RSI)
Description: The Reflux Symptom Index (RSI) is a validated questionnaire consisting of 9 statements to be ranked on a scale of 0-5 (0=no problem, 5=severe problem). RSI scores can range from 0 to 45, with higher scores correlated with more reflux symptoms.
Time Frame: baseline, 8 weeks
Population: There was no 8 week RSI score for the participant who withdrew from the amitriptyline arm so the change in score could not be calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 2 | 3
score on a scale | -2 (1.41) | -1.67 (2.08)

2. Secondary Outcome: Change in the Score on the Voice Handicap Index-10 (VHI-10)
Description: The Voice Handicap Index-10 (VHI-10) is a 10-question scale rated from 0-4 that addresses effects on quality of life from voice disorders (0=never, 1=almost never, 2=sometimes, 3=almost always, 4=always). VHI-10 scores can range from 0 to 40, with lower scores correlated with a higher quality of life related to voice disorders.
Time Frame: baseline, 8 weeks
Population: There was no 8 week VHI-10 score for the participant who withdrew from the amitriptyline arm so the change in score could not be calculated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale | 8.0 (11.31) | 2.67 (4.04)

3. Secondary Outcome: Change in the Score on the Cough Severity Index (CSI)
Description: The Cough Severity Index is a validated 10 item questionnaire to quantify a patient's symptoms associated with upper airway chronic cough. The 4 point Likert scale for each of the 10 items is 0 to 4 where 0 = Never, 1 = Almost never, 2 = Sometimes, 3 = Almost always, 4 = Always. Scores can range from 0 to 40 and higher scores reflect more coughing.
Time Frame: baseline, 8 weeks
Population: There was no 8 week CSI score for the participant who withdrew from the amitriptyline arm so the change in score could not be calculated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale | 10 (14.14) | 3.67 (5.51)

4. Secondary Outcome: Change in Throat Pain or Burning
Description: Participants will be asked to rate the severity of their "throat pain or burning" on a scale from 0 (no problem) to 5 (severe). Higher scores are correlated with more throat pain/burning.
Time Frame: baseline, 8 weeks
Population: There was no 8 week assessment of throat pain/burning for the participant who withdrew from the amitriptyline arm, so the change in score could not be calculated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale | 2.0 (2.83) | -1.33 (1.53)

5. Secondary Outcome: Change in Pain When Swallowing
Description: Participants were asked to rate their pain when swallowing on a scale of 0=none to 5= severe pain.
Time Frame: baseline, 8 weeks
Population: There was no 8 week assessment of pain while swallowing for the participant who withdrew from the amitriptyline arm, so the change in score could not be calculated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale | 1.0 (4.24) | 0.33 (1.53)

6. Secondary Outcome: Subjective Improvement of Laryngitis Symptoms
Description: Patients will subjectively rate improvement of symptoms on an ordinal 10-point scale where 0=no improvement and 10=significant improvement.
Time Frame: 8 weeks
Population: There was no 8 week assessment of subjective assessment of laryngitis symptoms for the participant who withdrew from the amitriptyline arm, so it could ot be reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale | 8.0 (0) | 2.0 (3.46)

7. Secondary Outcome: Number of Participants Who Dropped Out of the Study Due to Side Effects
Description: The number of patients who report they did not continue with study participation due to side effects, will be obtained from study logs.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Amitriptyline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amitriptyline (N=3) | Placebo (N=3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Arm weakness (General disorders) | 1 (1) | 0 (0)
Facial weakness (General disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lack of energy (General disorders) | 0 (0) | 1 (1)
Sleepy (General disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Funding was not obtained so the study could not be continued after the Covid pause.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT02552225/Prot_SAP_000.pdf